CLINICAL TRIAL: NCT03872960
Title: A Randomised Trial of Expedited Transfer to a Cardiac Arrest Centre for Non-ST Elevation Out-of-hospital Cardiac Arrest
Acronym: ARREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other); London School of Hygiene and Tropical Medicine (Other); Barts & The London NHS Trust (Other); King's College Hospital NHS Trust (Other); Imperial College Healthcare NHS Trust (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Royal Free Hospital NHS Foundation Trust (Other); St George's University Hospitals NHS Foundation Trust (Other); London Ambulance Service NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MJKTUAR; ISRCTN96585404 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2019-03-08; First posted 2019-03-13 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: cardiac arrest; pre-hospital care; strategy trial
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm: Expedited transfer to a CAC (Experimental): The intervention arm consists of activation of the pre-hospital triaging system currently in place for post-arrest STE patients. This involves pre-alert of the CAC and strategic delivery of the patient to the catheter laboratory (24 hours a day, 7 days a week). Patients will receive definitive post-resuscitation care: intubation and ventilation, where necessary, targeted temperature management, and goal directed therapies including evaluation and identification of underlying cause of arrest with access to immediate reperfusion if necessary. Prognostication will occur no earlier than 72 hours post-cardiac arrest to prevent premature withdrawal of life-sustaining treatment. Transfer times estimated from the 40-patient pilot are anticipated to be 100 minutes (median; IQR 75 to 113) from time of arrest to the designated centre.
  Interventions: Procedure: Transfer to cardiac arrest centre
- Control Arm: Current standard of care (No Intervention): The control arm comprises the current standard of pre-hospital advanced life support (ALS) care management for patients with ROSC following cardiac arrest of suspected cardiac aetiology. The patient is conveyed to the geographically closest emergency department. Management thereafter will be as per standard hospital protocols however as in the intervention arm, prognostication is to be delayed in trial patients until at least 72 hours post arrest.

INTERVENTIONS:
Procedure: Transfer to cardiac arrest centre — Patients in the intervention arm will be taken directly to a the catheter lab of a heart attack centre.
  Arms: Intervention Arm: Expedited transfer to a CAC

SUMMARY:
The aim of ARREST is to determine the best post-resuscitation care pathway for out of hospital cardiac arrest patients without ST-segment elevation. The investigators propose that changes to emergency management comprising expedited delivery to a specialist heart attack centre with organised post-cardiac arrest care including immediate access to reperfusion therapy will reduce mortality in patients without STE compared to the current standard of care, which comprises protracted pre-hospital management of the patient without definitive care plan and delivery to geographically closest hospital.

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest (OHCA) is a global public health issue. There are 60,000 cardiac arrests per year in the United Kingdom (UK), of which resuscitation is attempted in just under half. Resuscitation attempts are successful in up to 30%. However, more than two thirds of patients who survive to hospital admission die before discharge. There is wide variation in both regional and inter-hospital survival rates from OHCA; this disparity is also present across London. This variation has been shown to be attributable to hospital infrastructure, resources and personnel rather than patient characteristics. Overall survival therefore remains poor, at 7%.

It is well known that the majority of OHCA are secondary to an acute cardiac ischaemic event. Coronary artery disease is responsible for more than 70% of OHCA of presumed cardiac cause, with acute occlusion demonstrated in 50% of consecutive patients taken for immediate coronary angiography (ICA). Early cardiopulmonary resuscitation (CPR) and defibrillation, with ICA and percutaneous coronary intervention (PCI) in a cardiac arrest centre (CAC), prevents re-arrest, preserves myocardial function and has been shown to improve post-arrest outcomes in ST-segment elevation (STE). The management of patients without STE however is controversial, with a delayed approach to intervention. Despite recently published data suggesting PCI in non-STE resulted in a two-fold increase in favourable outcome, randomised data are lacking. Emergent reperfusion therapies come with a weak recommendation from the International Liaison Committee on Resuscitation (ILCOR), and a Class IIa recommendation by the American Heart Association (AHA) and European Society of Cardiology (ESC), if there is a high suspicion of ongoing infarction.

The European Association of Percutaneous Cardiovascular Interventions (EAPCI) recommends a prior rule-out of non-cardiac cause in the emergency department followed by coronary angiography within 2 hours. It remains unclear if time-critical, definitive hospital based management of the post-arrest patient without STE in a specialist centre improves outcomes, and there has been variable uptake of this strategy both pre-hospital and amongst the interventional cardiology community.

There is an urgent need for a randomised controlled trial examining the benefits of early delivery of post-cardiac arrest care in specialist centres, specifically in the absence of STE. Post-arrest care is time-critical, requires a multi-disciplinary approach and may be more optimally delivered in centres with greater provider experience. ILCOR and the EAPCI state that randomised trials are essential in this population to determine if timely delivery by the ambulance services to a CAC with organised postcardiac arrest care including immediate access to reperfusion therapy improves survival. There are no randomised trials and only indirect evidence that CAC and systems of care may be effective and only two observational studies examining the role of immediate ICA±PCI in the absence of STE. This is an important and topical question as there is a drive to regionalise care for all patients into CACs.

To address this, ARREST will enroll 860 OHCA patients with ROSC to a randomised clinical trial. Each arm of the trial will include 430 patients.

The two arms are as follows:

Intervention Arm: Direct to CAC The intervention arm consists of activation of the pre-hospital triaging system currently in place for post-arrest STE patients. This involves pre-alert of the CAC and strategic delivery of the patient to the catheter laboratory (24 hours a day, 7 days a week). Patients will receive definitive post-resuscitation care: intubation and ventilation, where necessary, targeted temperature management, and goal directed therapies including evaluation and identification of underlying cause of arrest with access to immediate reperfusion if necessary. Prognostication will occur no earlier than 72 hours post-cardiac arrest to prevent premature withdrawal of life-sustaining treatment. Transfer times estimated from the 40-patient pilot are anticipated to be 100 minutes (median; IQR 75 to 113) from time of arrest to the designated centre.

Control Arm: Standard of Care The control arm comprises the current standard of pre-hospital advanced life support (ALS) care management for patients with ROSC following cardiac arrest of suspected cardiac aetiology. The patient is conveyed to the geographically closest emergency department. Management thereafter will be as per standard hospital protocols however as in the intervention arm, prognostication is to be delayed in trial patients until at least 72 hours post arrest.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest (OHCA)
* Return of spontaneous circulation (ROSC)
* Age 18 or over (known or presumed)

Exclusion Criteria:

* Criteria for ST-elevation myocardial infarction on 12-Lead electrocardiogram (ECG)
* Do Not Attempt Resuscitation (DNAR) Order
* Cardiac arrest suffered after care pathway set and patient en route
* Suspected pregnancy
* Presumed non-cardiac cause (for example; trauma, drowning, suicide, drug overdose)
* Presumed significant trauma/injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 862 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 30 days after randomisation

SECONDARY OUTCOMES:
Cerebral performance category score | Discharge (capped at 30 days)
  Neurological status assessed using the cerebral performance category (ranked scale from 1 to 5 with 1 being the best outcome and 5 the worse outcome)
Modified Rankin Score | Discharge (capped at 30 days)
  Neurological status assessed using the modified Ranking Score (ranked scale from 0 to 6 with 0 being the better outcome and 6 the worse outcome).
Cerebral performance category score | 3 months after randomisation
  Neurological assessed using the cerebral performance category (ranked scale from 1 to 5 with 1 being the best outcome and 5 the worse outcome)
Modified Rankin Score | 3 months after randomisation
  Neurological status assessed using the modified Ranking Score (ranked scale from 0 to 6 with 0 being the better outcome and 6 the worse outcome).
All-cause mortality | 3 months after randomisation
All-cause mortality | 6 months after randomisation
All-cause mortality | 12 months after randomisation
Patient's quality of life | Discharge (capped at 30 days)
  Assessed using the EuroQol-5 Dimension-5 Level (EQ-5D-5L) standardised survey

CONTACTS AND LOCATIONS:
Overall Officials: Simon Redwood, MBBS, PhD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (22):
- United Kingdom (22):
  - Dartford and Gravesham NHS Trust, Dartford
  - Barts Health NHS Trust, London
  - BHR University Hospitals NHS Trust, London
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - Croydon Health Services NHS Trust, London
  - Epsom and St Helier University Hospitals NHS Trust, London
  - Guy's and St Thomas' NHS FT, London
  - Hillingdon Hospitals NHS Trust, London
  - Homerton University Hospital NHS Trust, London
  - Imperial College Healthcare NHS Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Kingston Hospital NHS FT, London
  - Lewisham & Greenwich NHS Trust, London
  - London Ambulance Service NHS Trust, London
  - London North West University Healthcare, London
  - North Middlesex University Hospital NHS Trust, London
  - Royal Brompton and Harefield NHS Trust, London
  - Royal Free London NHS Foundation Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Surrey and Sussex Healthcare NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - West Hertfordshire Hospitals NHS Trust, Watford

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Patterson T, Perkins A, Perkins GD, Clayton T, Evans R, Nguyen H, Wilson K, Whitbread M, Hughes J, Fothergill RT, Nevett J, Mosweu I, McCrone P, Dalby M, Rakhit R, MacCarthy P, Perera D, Nolan JP, Redwood SR. Rationale and design of: A Randomized tRial of Expedited transfer to a cardiac arrest center for non-ST elevation out-of-hospital cardiac arrest: The ARREST randomized controlled trial. Am Heart J. 2018 Oct;204:92-101. doi: 10.1016/j.ahj.2018.06.016. Epub 2018 Aug 6. PMID 30092413
- [Result] Patterson T, Perkins GD, Perkins A, Clayton T, Evans R, Dodd M, Robertson S, Wilson K, Mellett-Smith A, Fothergill RT, McCrone P, Dalby M, MacCarthy P, Firoozi S, Malik I, Rakhit R, Jain A, Nolan JP, Redwood SR; ARREST trial collaborators. Expedited transfer to a cardiac arrest centre for non-ST-elevation out-of-hospital cardiac arrest (ARREST): a UK prospective, multicentre, parallel, randomised clinical trial. Lancet. 2023 Oct 14;402(10410):1329-1337. doi: 10.1016/S0140-6736(23)01351-X. Epub 2023 Aug 27. PMID 37647928

DOCUMENTS (1):
  • Study Protocol (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT03872960/Prot_000.pdf